CLINICAL TRIAL: NCT05062525
Title: Immune Response to COVID-19 Vaccine in Immunotherapy (IO) and Non-IO Treated Cancer Patients
Acronym: VIVACIOUS
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: VIVACIOUS; 21-5797 (Other: REB ID)
Record Dates: First submitted 2021-09-29; First posted 2021-09-30 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; Cancer
Keywords: COVID-19 Vaccine
MeSH Terms: conditions — COVID-19; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immunotherapy
- Non-Immunotherapy

SUMMARY:
Evaluation of antibody response against SARS-CoV-2 vaccination in patients treated with IO-treatment, in comparison with antibody titers in patients treated with non-IO treatment.

DETAILED DESCRIPTION:
Blood samples will be analyzed to determine the magnitude of SARS-CoV-2 immunity in cancer patients treated with immunotherapy by quantifying antibodies and other tumor or blood-based biomarkers against SARS-CoV-2 epitopes following vaccination. We will also explore for potential development of autoantibodies and other blood-based biomarkers, following SARS-CoV-2 vaccination, and their correlation with clinical manifestation of IO related immune-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with solid malignancies treated with either IO or non-IO treatment.
2. All categories of IO treatment allowed (immune-checkpoint inhibitors, bi-specific T cell engagers, cytokine agonists and others), as well as all categories of non-IO treatment (such as chemotherapy and targeted therapies). These can be given as part of standard of care or within participation in a clinical trial.
3. Patients are allowed to have any of the approved vaccines in Canada, such as Pfizer, Moderna, AstraZeneca or their approved combinations.
4. Patients must receive all appropriate doses of SARS-CoV-2 vaccination, as dictated by the respective vaccine schedules.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid malignancies treated with either immunotherapy or non-immunotherapy treatment who have received the SARS-CoV-2 vaccination.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Concentration of SARS-CoV-2 antibodies | 15 months
Number of immune-related adverse events | 15 months

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada